CLINICAL TRIAL: NCT00704223
Title: Observational Study on Safety and Efficacy in Subjects Using NovoMix® 70 (Biphasic Insulin Aspart) for Treatment of Type 2 Diabetes Mellitus
Brief Title: Observational Study to Evaluate the Safety and Efficacy of NovoMix® 70 in Type 2 Diabetes
Acronym: INTENSIV
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: BIASP-3576
Record Dates: First submitted 2008-06-20; First posted 2008-06-24 (Estimated); Last update posted 2014-06-24 (Estimated); Status verified 2014-06

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — insulin aspart, insulin aspart protamine drug combination 30:70

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood sample
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- A
  Interventions: Drug: biphasic insulin aspart

INTERVENTIONS:
Drug: biphasic insulin aspart — Start dose and frequency to prescribed by the physician as a result of a normal clinical evaluation
  Other Names: NovoMix® 70

SUMMARY:
This study is conducted in Europe. The aim of this observational study is to evaluate the incidence of adverse events while using NovoMix® 70 under normal clinical practice conditions in Austria.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes
* HbA1c over 7%
* No contraindication with NovoMix® 70

Exclusion Criteria:

* Type 1 diabetes
* Subjects participating in a clinical trial or another observational study
* Subjects under previous basis-bolus insulin therapy
* Women who are pregnant, breast feeding and women of child bearing capacity who are not using any reliable contraceptive method

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male and female above 18 years with type 2 diabetes
Sampling Method: Probability Sample
Enrollment: 619 (Actual)
Dates: Start 2008-05; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
number of major and minor hypoglycaemic events and adverse events | 3 months

SECONDARY OUTCOMES:
HbA1c | 3 months
PPBG | 3 months
FBG | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Vienna, Austria

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com